CLINICAL TRIAL: NCT00975429
Title: Vascular-Targeted Photodynamic Therapy Using WST11 in Patients With Localized Prostate Cancer
Brief Title: Study Using WST11 in Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN902 PCM203
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: Prostatic Disease; Genital neoplasm, male; Urogenital neoplasm; Genital disease,male; Male urogenital disease; Neoplasms; Neoplasm by site; Prostatic neoplasm; Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Carcinoma | interventions — padeliporfin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WST11 - 4mg (TOOKAD® Soluble) (Experimental): 4mg/kg Treatment with WST11-mediated VTP
  Interventions: Drug: WST11
- WST11 - 6mg (Experimental): 6mg/kg Treatment with WST11-mediated VTP
  Interventions: Drug: WST11

INTERVENTIONS:
Drug: WST11 — The WST11-mediated VTP procedure will consist of a single IV administration of WST11 at a dose of 4mg/kg using a 753nm laser light at a fixed power (150mW/cm or 200mW/cm or 250mW/cm) and light energy (200J/cm or 300J/cm) delivered through transperineal interstitial optical fibers. The fibers are introduced into transparent needles that are positioned in the prostate under ultra sound image guidance. The tumour location is established using transrectal biopsy and MR imaging. The number of fibers and the total light energy will be adapted to each patient based on a treatment planning proposed by treatment planning group.
  Other Names: Treatment with WST11-mediated VTP
  Arms: WST11 - 4mg (TOOKAD® Soluble)
Drug: WST11 — The WST11-mediated VTP procedure will consist of a single IV administration of WST11 at a dose of 6mg/kg in patients using a 753nm laser light at a fixed power (150mW/cm or 200mW/cm or 250mW/cm ) and light energy (200J/cm or 300J/cm) delivered through transperineal interstitial optical fibers. The fibers are introduced into transparent needles that are positioned in the prostate under ultra sound image guidance. The tumour location is established using transrectal biopsy and MR imaging. The number of fibers and the total light energy will be adapted to each patient based on a treatment planning proposed by treatment planning group.
  Other Names: Treatment with WST11-mediated VTP
  Arms: WST11 - 6mg

SUMMARY:
The aim of this trial is to determine the optimal treatment conditions to achieve prostate cancer tumour ablation and to assess the effects of WST11-mediated Vascular-Targeted Photodynamic therapy (VTP) treatment in patients with localized prostate cancer.

The secondary objectives are to assess the safety and quality of life following WST11-mediated VTP treatment,to assess the effects,safety and quality of life following a second WST11-mediated VTP treatment; and to explore optimisation techniques to reduce the duration of the VTP procedure.

DETAILED DESCRIPTION:
This trial is designed as a multicentre, phase II, open-labeled, multi-arm, single intravenous (IV) dose study. The patient is to receive general anesthesia. WST11-mediated VTP will consist of the combination of a single IV administration of WST11 at doses of 4 or 6 mg/kg using 753nm laser light at a fixed power (150 mW/cm or 200 mW/cm or 250 mW/cm ) and light energy (200 J/cm or 300J/cm) delivered through transperineal interstitial optical fibers. The fibers are introduced into transparent needles that are positioned in the prostate under ultra sound guidance. The tumour location is established using transrectal biopsy and MR imaging. The number of fibers and the total light energy will be adapted to each patient based on a treatment planning proposed by treatment planning group.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years of age;
* Diagnosed with prostate cancer and eligible for active surveillance;
* No prior treatment for prostate cancer;
* Prostate Cancer Stage up to cT2b - N0/Nx - M0/Mx (rT2c and pT2c are acceptable)
* Gleason score ≤ 3+3 For patients characterized with prostate mapping (transperineal template guided biopsy at 5mm intervals) a secondary pattern 4 is acceptable provided that it is not present in more than 3 cores from each side of the prostate and is no more than 3 mm cancer core length.
* PSA < 10 ng/mL;
* Signed Informed Consent Form.

Exclusion Criteria:

* Any condition or history of illness or surgery that, in the opinion of the investigator and/or the Sponsor, might confound the results of the study or pose additional risks to the patient.
* All patients whose current pre-operative cardiac evaluation does not show their fitness for a procedure requiring general anesthesia;
* Patients with a prior history of viral or alcoholic hepatitis, and other patients felt to be at risk for hepatotoxicity including concomitant use of potentially hepatotoxic medications or dietary supplements;
* Patients with a history of inflammatory bowel disease or other factors which may increase the risk of fistula formation;
* Men who have received any hormonal manipulation (excluding 5-alpha reductase inhibitors) or androgen supplements within the previous 6 months;
* Men previously treated by radiation therapy (external therapy or brachytherapy) or chemotherapy or any therapy for prostate cancer;
* Men who have received or are receiving chemotherapy for prostate carcinoma or other significant cancer;
* Men who have undergone previous TURP (trans-urethral resection of the prostate);
* Men who are currently receiving any medications having potential photosensitizing effects (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics and griseofulvin).
* Men who are receiving anticoagulant drugs (e.g.: coumadin, warfarin).
* Patient who stopped long term treatment of acetylsalicylic acid (aspirin) or other anti platelets agents less than 15 days before the procedure;
* Patient suspected of Disseminated Intravascular Coagulation (DIC) as defined by the presence of three out of the five following criteria: platelets <LLN, PT >ULN, aPTT >ULN, fibrinogen<LLN, D-Dimer >ULN
* History of non compliance with medical therapy and medical recommendations or an unwillingness or inability to complete patient self-administered questionnaires;
* Participation in a clinical study or receipt of an investigational treatment within the past 3 months;
* A history of porphyria;
* A history of sun hypersensitivity or photosensitive dermatitis;
* Renal disorders (blood creatinine > 1.5 x ULN) or known post mictional residue > 150cc
* Hepatic disorders (transaminases > ULN, bilirubin > ULN,). In case of slight abnormalities, another exam should be performed. If the results are within normal ranges, then the patient can be included;
* Hematological disorders (white cells < 2500/mm3, neutrophils < 1500/mm3, platelets < 140.000/mm3, Hb < 8 g/dL);
* Patient with contra-indication to MRI (such as pace maker, metal prosthesis, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Negative biopsy in the treated lobes | Month 6

SECONDARY OUTCOMES:
Serum PSA levels and PSA changes after treatment compared to baseline. | Month 1, Month 3 & Month 6
Volume of hypoperfusion area shown by dynamic gadolinium MRI. | Day 7, Month 6
Adverse events, ECG (12-lead),vital signs,clinical laboratory evaluations, physical examination. | Screening-Month 6
Quality of life IPSS; IIEF | Month 1, Month 3 & Month 6
Optimisation of the procedure | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, Professor, Principal Investigator — University College London Hospital (UCLH); Gordon MUIR, MD, Principal Investigator — Kings College Hospital (KCH); Neil BARBER, MD, Principal Investigator — Frimley Park Hospital NHS Trust; Michel de Wildt, MD, Principal Investigator — Catharina Ziekenhuis; Abdel-Rahmène AZZOUZI, Professor, Principal Investigator — Centre Hospitalier Unniversitaire Angers(CHU); Eric BARRET, MD, Principal Investigator — Institut Mutualiste Montsouris (IMM); Arnauld VILLERS, Professor, Principal Investigator — Hôpital Claude-Huriez
Locations (7):
- France (3):
  - Centre Hospitalier Universitaire (CHU), Angers
  - Hôpital Claude Huriez, Lille
  - Institut Mutualiste Montsouris(IMM), Paris
- Catharina Ziekenhuis, Eindhoven, Netherlands
- United Kingdom (3):
  - Frimley Park Hospital NHS Trust, Frimley
  - Kings College Hospital (KCH), London
  - University College London Hospital (UCLH), London

REFERENCES:
- [Result] Azzouzi AR, Barret E, Moore CM, Villers A, Allen C, Scherz A, Muir G, de Wildt M, Barber NJ, Lebdai S, Emberton M. TOOKAD((R)) Soluble vascular-targeted photodynamic (VTP) therapy: determination of optimal treatment conditions and assessment of effects in patients with localised prostate cancer. BJU Int. 2013 Oct;112(6):766-74. doi: 10.1111/bju.12265. PMID 24028764
- [Derived] Azzouzi AR, Lebdai S, Benzaghou F, Stief C. Vascular-targeted photodynamic therapy with TOOKAD(R) Soluble in localized prostate cancer: standardization of the procedure. World J Urol. 2015 Jul;33(7):937-44. doi: 10.1007/s00345-015-1535-2. Epub 2015 Mar 19. PMID 25786708
- [Derived] Azzouzi AR, Barret E, Bennet J, Moore C, Taneja S, Muir G, Villers A, Coleman J, Allen C, Scherz A, Emberton M. TOOKAD(R) Soluble focal therapy: pooled analysis of three phase II studies assessing the minimally invasive ablation of localized prostate cancer. World J Urol. 2015 Jul;33(7):945-53. doi: 10.1007/s00345-015-1505-8. Epub 2015 Feb 25. PMID 25712310
- [Derived] Lebdai S, Villers A, Barret E, Nedelcu C, Bigot P, Azzouzi AR. Feasibility, safety, and efficacy of salvage radical prostatectomy after Tookad(R) Soluble focal treatment for localized prostate cancer. World J Urol. 2015 Jul;33(7):965-71. doi: 10.1007/s00345-015-1493-8. Epub 2015 Jan 23. PMID 25614256